CLINICAL TRIAL: NCT07401056
Title: The Effect of Preoperative Structured Exercise Programme on Postoperative Pain Severity, Recovery Level, Discharge Time and Quality of Life in Patients With Non-Small Cell Lung Cancer: Randomised Controlled Study
Brief Title: Preoperative Structured Exercise Programme on Patients With Non-Small Cell Lung Cancer
Acronym: READY-LUNG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Burcu Duluklu, Asst. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HAE24/90
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: exercise; discharge; lung cancer; pain; prehabilitation; quality of life; recovery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity; Lung Neoplasms; Pain | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Prehabilitation (Structured Preoperative Exercise Programme)
  Interventions: Other: Prehabilitation (Structured Preoperative Exercise Programme)
- Control Group (No Intervention): Control: Partients in this arm will receive standard preoperative care without a structured exercise programme. Study-related data will be collected from patients admitted to the hospital at the end of the two-week preoperative period in accordance with the study protocol. In this regard, the measurements to be taken in the study will include: (1) Pain severity: At 6, 12, 24 and 48 hours after surgery; (2) Surgical recovery level: On the third and seventh days after surgery; (3) Quality of life: On the first day before surgery and on the seventh day after surgery. (4) In addition, patients' LOSs will be recorded.

INTERVENTIONS:
Other: Prehabilitation (Structured Preoperative Exercise Programme) — Participants in this arm will receive a structured preoperative exercise programme starting two weeks before surgery. The programme includes moderate-intensity walking for at least 30 minutes 5 days per week, deep breathing and coughing exercises four times daily, and hourly incentive spirometry exercises while awake. Participants will record daily adherence to the exercise programme, and compliance will be monitored through daily telephone follow-up by the researcher. Study-related data will be collected from patients admitted to the hospital at the end of the two-week preoperative period in accordance with the study protocol. In this regard, the measurements to be taken in the study will include: (1) Pain severity: At 6, 12, 24 and 48 hours after surgery; (2) Surgical recovery level: On the third and seventh days after surgery; (3) Quality of life: On the first day before surgery and on the seventh day after surgery. (4) In addition, patients' LOSs will be recorded.
  Arms: Intervention Group

SUMMARY:
INTRODUCTION: Lung cancer is among the leading cancers, and surgery has a major role in treatment. Patients diagnosed with Non-Small Cell Lung Cancer (NSCLC) who are eligible for surgical treatment have a high risk of experiencing postoperative complications. Therefore, in recent years, the concept of prehabilitation has begun to gain importance. Within the scope of prehabilitation practices, patients are provided with programmes that include aerobic exercises and breathing exercises in the preoperative period.

AIM: This study aims to evaluate the effects of a structured exercise programme, including aerobic exercises and breathing exercises in the preoperative period, on postoperative pain severity, surgical recovery level, length of hospital stays (LOS), and quality of life (QoL) in patients diagnosed with NSCLC and planned for surgical treatment.

METHODS: The research is an experimental, parallel group-randomised controlled trial to be conducted with 62 participants followed in the Thoracic Surgery Outpatient Clinic of Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital and scheduled for surgery due to NSCLC. Patients will be equally assigned to the intervention and control groups using the block randomization method. In the intervention group, in the preoperative period, for two weeks and five days per week, at least 30 minutes of walking per day will be performed; in addition, for two weeks before surgery, throughout the entire week, during waking hours, 10 repetitions with incentive spirometer every hour, and daily four sessions of deep breathing & coughing exercises will be performed as breathing exercises. In the control group, routine preoperative clinical procedures will be applied. In the postoperative period, pain severity, surgical recovery level, LOS, and QoL will be compared between the two groups. Data will be collected face-to-face by the researcher using the "Descriptive Characteristics Form", "EQ-5D-5L Quality of Life Scale", "Numeric Rating Scale (NRS)", and "Surgical Recovery Scale". Data on the length of hospital stay will be obtained from patient files. The data will be analysed using parametric and/or nonparametric tests through the SPSS.

CONCLUSION: The findings of the study are expected to contribute to strengthening holistic care approaches for the preoperative period in surgical nursing practices and to improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. Ownership of a smartphone capable of tracking daily walking time.
3. Diagnosis of primary non-small cell lung cancer.
4. ASA (American Society of Anesthesiologists) classification I, II, or III.
5. Follow-up and treatment provided by the same surgical team.
6. No physical or cognitive impairment that would hinder participation in the study.

Exclusion Criteria

1. Diagnosis of recurrent lung cancer.
2. Previous radiotherapy treatment prior to surgery.
3. Any condition preventing walking or exercise (orthopedic, neurological, cardiovascular, metastatic, etc.).
4. Diagnosis of additional respiratory system disease such as COPD, asthma, or emphysema preventing breathing exercises.
5. Inability to complete the two-week structured exercise programme due to surgery being scheduled earlier or later than planned.
6. Complications resulting in prolonged (>24 hours) intensive care unit stay after surgery.
7. Inability to discontinue or continue the structured exercise programme at any stage.
8. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (EQ-5D-5L) | Change from baseline scores on the 7th postoperative day.
  The EQ-5D-5L is a self-reported questionnaire assessing five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, mild problems, moderate problems, severe problems, and extreme problems. The questionnaire also includes a Visual Analog Scale (VAS) ranging from 0 (worst health) to 100 (best health) for participants to rate their current health status. Higher scores indicate better health.
Postoperative Pain Intensity (Numeric Rating Scale, NRS) | Change from baseline scores on the 48 hours postoperatively.
  The NRS is an 11-point scale (0-10) used to assess pain intensity, where 0 indicates no pain and 10 indicates the worst possible pain. Patients rate their pain at each time point, and the average of the measurements will be used to assess postoperative pain. The NRS is validated for adults, including elderly patients and those with mild-to-moderate cognitive impairment.
Postoperative Surgical Recovery (Surgical Recovery Scale) | Change from baseline scores on the 7th postoperative day.
  The Surgical Recovery Scale is a 13-item questionnaire assessing two sub-dimensions: "Impact on energy" and "Impact on daily activities." Items are scored using 6-point Likert scales, with higher scores indicating better recovery. The total score ranges from 8 to 73. This scale is validated with a Cronbach's α of 0.93.

SECONDARY OUTCOMES:
Length of Hospital Stay | Approximately the seventh day.
  Patients' discharge time will be recorded and compared in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Duluklu, Asst. Prof., Principal Investigator — Hacettepe University, Faculty of Nursing, Surgical Nursing Department
Locations (1):
- Hacettepe University, Ankara, Altındağ 06230, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz B, Yayla A. Validity and Reliability Study of the Turkish Version of the Surgical Recovery Scale. J Perianesth Nurs. 2025 Oct;40(5):1281-1289. doi: 10.1016/j.jopan.2025.01.023. Epub 2025 Jun 20. PMID 40542811
- [Result] Machado P, Pimenta S, Garcia AL, Nogueira T, Silva S, Dos Santos CL, Martins MV, Canha A, Oliveiros B, Martins RA, Cruz J. Effect of Preoperative Home-Based Exercise Training on Quality of Life After Lung Cancer Surgery: A Multicenter Randomized Controlled Trial. Ann Surg Oncol. 2024 Feb;31(2):847-859. doi: 10.1245/s10434-023-14503-2. Epub 2023 Nov 7. PMID 37934383
- [Result] Jiao M, Liang H, Zhang M. Effect of exercise on postoperative recovery of patients with non-small cell lung cancer: a systematic review and meta-analysis. Discov Oncol. 2024 Jun 17;15(1):230. doi: 10.1007/s12672-024-01079-w. PMID 38884823
- See also: EQ-5D-5L Quality of Life Scale — https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-y-5l/